CLINICAL TRIAL: NCT06677294
Title: The Effects of Intrauterine Interventions During Placenta Removal on Pain, Perception of Traumatic Birth, and Early Postpartum Health Indicators in Women
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Deniz Akyıldız, Assoc. Prof. Dr., Kahramanmaras Sutcu Imam University
Other Study IDs: Placenta Removal Interventions
Record Dates: First submitted 2024-09-23; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2023-09

CONDITIONS: Placenta, Retained
MeSH Terms: conditions — Placenta, Retained

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: while those who did not undergo such interventions were placed in the control group
  Interventions: Procedure: Placenta remove
- Case: In the study, women who underwent intrauterine interventions during the third stage of labor for placental removal were included in the case group (n=32), while those who did not undergo such interventions were placed in the control group (n=32). Manual placental removal (hallas) and the cleaning of the uterine cavity using the hand or gauze/sponge (wrapped around the hand or using an over-clamp) after placental expulsion were considered intrauterine interventions
  Interventions: Procedure: Placenta remove

INTERVENTIONS:
Procedure: Placenta remove — This is an observational study. No intervention was performed

SUMMARY:
A prospective cohort study was conducted with 64 women who had vaginal deliveries at Adana City Training and Research Hospital between October 2023 and May 2024. Women who received intrauterine interventions during the third stage of labor formed the case group (n=32), and those who did not formed the control group (n=32). Data were collected using the Pregnant Information Form, Labor Observation Form, Early Postpartum Period Follow-up Form, Visual Analog Scale (VAS), and Traumatic Birth Perception Scale (TBPS). Findings were determined through regular monitoring and follow-ups during the first 24 hours postpartum.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria required participants to be 18 years or older, to have delivered at term (38-40 weeks), to have had a vaginal delivery, and to have a singleton pregnancy. Additionally, participants must not have been using analgesic medications, must not have had hypertension or preeclampsia, and must not have experienced atony in a previous pregnancy. Participants also needed to be free from infections, placental anomalies, genital lesions, or coagulation disorders, and they had to agree to participate in the study

Exclusion Criteria:

Exclusion criteria included women who experienced a difficult labor or whose delivery involved the use of forceps or vacuum assistance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria required participants to be 18 years or older, to have delivered at term (38-40 weeks), to have had a vaginal delivery, and to have a singleton pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Women's pain levels | VAS scores were recorded at 10 minutes, 30 minutes, 1 hour, 12 hours, and 24 hours postpartum
  The Visual Analog Scale (VAS) was used to assess pain levels in this study. The VAS is a continuous scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst possible pain." Higher scores on the VAS indicate a worse outcome, as they reflect greater levels of reported pain.
Traumatic Birth Perception | At 24 hours postpartum
  The Traumatic Birth Perception Scale (TBPS) was developed to measure the perception of traumatic birth in women and consists of 13 items within a single subdimension. There are no reverse-scored items in the scale, and each item is rated on a scale of 0 to 10. The lowest possible score is 0, and the highest possible score is 130. The total score reflects the level of traumatic birth perception, with higher scores indicating a higher perception of trauma related to the birth experience.
Early postpartum health characteristics | 10th minute, 15th minute, 20th minute, 30th minute, 45th minute, 60th minute, 90th minute, 2nd hour, 3rd hour, 4th hour, 5th hour, 6th hour, 12th hour, 18th hour and 24th hour

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No